CLINICAL TRIAL: NCT06043648
Title: The Role of Continuous Endotracheal Tube Cuff Pressure Monitoring With a Simple Method in the Incidence of Endotracheal Tube-related Complications
Brief Title: Continuous Endotracheal Tube Cuff Pressure Monitoring
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Demet Laflı Tunay, Principal Investigator, Cukurova University
Other Study IDs: CUFFP
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Complications Related to Endotracheal Intubation
Keywords: cuffed endotracheal tube, intracuff pressure, pressure transducer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Constant monitoring: Intracuff pressure was monitored continuously throughout the surgery using the transducer of the invasive pressure monitoring device in patients undergoing elective non-head-neck surgical procedures under general anesthesia and orally intubated with a cuffed endotracheal tube.
  Interventions: Device: Endotracheal tube cuff pressure monitoring
- Intermittent monitoring: Intracuff pressure was monitored intermittently throughout the surgery using an analogue manometer in patients undergoing elective non-head-neck surgical procedures under general anesthesia and orally intubated with a cuffed endotracheal tube.
- None monitoring: After endotracheal intubation with a cuffed endotracheal tube, the cuff was inflated by the anesthesia provider using sealing pressure technique which involves slow inflation of the cuff until there is no audible gas leak while holding continuous positive airway pressure of 20 cmH2O with the head and neck in the neutral position. No other intracuff pressure monitoring or measurement was performed throughout the operation.

INTERVENTIONS:
Device: Endotracheal tube cuff pressure monitoring — The endotracheal tube cuff pressure was continuously monitored using a transducer from a standard invasive pressure monitoring device that is routinely used to measure arterial or central venous pressure.
  Groups: Constant monitoring

SUMMARY:
Tracheal tube cuff pressure in the range of 20 to 30 cmH2O is considered safe, but it is quite common to encounter cuff pressure outside this range in patients with tracheal intubation. Moreover, objective cuff pressure measurement and monitoring are not routinely applied, especially in general anesthesia practice. Overinflation of the cuff can potentially impair tracheal mucosal blood flow. This may lead to various tracheal injuries such as mucosal inflammation, mucosal ischemia, tracheal ulceration, tracheal stenosis, tracheoesophageal fistula, and tracheal rupture. Conversely, inadequate cuff inflation can lead to inadequate ventilation and microaspiration. The importance of routine cuff pressure measurement and pressure adjustment to keep the pressure in the desired range is emphasized in preventing such side effects in intubated patients. Despite this recommendation for routine intracuff pressure measurement, the methods used to measure and monitor cuff pressure vary from subjective estimation techniques to objective measurements, and there is a lack of specific protocols and documents in the current literature. For this purpose, in this study, it was aimed to perform continuous cuff pressure measurement monitoring using the transducer of the invasive pressure monitoring device, which is routinely used in arterial or central venous pressure monitoring, and to test the effectiveness of this method in reducing cuff-related complications including sore throat, hoarseness, and dysphagia compared to the intermittent monitoring method.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age adult patients
* Elective non-head-neck surgical procedures under nitrous oxide (N2O)-free general anesthesia
* Patients orally intubated with a cuffed endotracheal tube facilitated by neuromuscular blockers
* Surgeries with neutral head-neck position

Exclusion Criteria:

* Emergency surgery
* Laparoscopic surgery
* Head and neck surgeries including nose, mouth, pharynx, larynx and throat
* Surgeries with non-supine patient position
* Patients with preoperative sore throat, cough, hoarseness or dysphagia, history of smoking, asthma or COPD, severe cardiovascular disease, inability to obtain consent, having any lesions detected in the pharynx or larynx during laryngoscopy
* Use of double lumen tracheal tube
* Use of a naso- or orogastric tube or any pharyngeal catheter
* Intraoperative nitrous oxide use
* Difficult intubation or repeated endotracheal intubation attempt
* Patients who strain during endotracheal extubation
* High PEEP (greater than 5 cmH2O) application

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for elective non-head-neck surgical procedures under N2O-free general anesthesia and orally intubated with a cuffed endotracheal tube facilitated by neuromuscular blockers.
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative sore throat | Postoperative 2 and 24 hours
  The incidence of endotracheal tube-related complication defined as sore throat during postoperative 2 and 24 hours.
Incidence of postoperative hoarseness | Postoperative 2 and 24 hours
  The incidence of endotracheal tube-related complication defined as hoarseness during postoperative 2 and 24 hours.
Incidence of postoperative dysphagia | Postoperative 2 and 24 hours
  The incidence of endotracheal tube-related complication defined as dysphagia during postoperative 2 and 24 hours.

SECONDARY OUTCOMES:
Identification of predictive factors related to endotracheal tube-related complications | During postoperative 24 hours
  Identification of patient and operative characteristics and mechanical ventilation related factors that influence ETT-related complications.

CONTACTS AND LOCATIONS:
Overall Officials: Demet Laflı Tunay, Dr., Principal Investigator — Çukurova University, Balcalı Hospital
Locations (1):
- Çukurova University; Faculty of Medicine, Adana, Sarıçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All data were anonymized by the local researcher. Therefore, data collection was pseudonymous and the patient's name did not appear on any case report form or other study document. All collected data were kept confidential. This study was conducted in accordance with the revision of the Declaration of Helsinki (2008). ICH-GCP was strictly adhered to.